CLINICAL TRIAL: NCT06876519
Title: Clinical Efficacy of Different Maxillary Sinus Floor Elevation Procedures Based on Maxillary Sinus Anatomy
Brief Title: Clinical Efficacy of Different Maxillary Sinus Floor Elevation Procedures
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital of Stomatology, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wang Jinming, Chief Physician, Hospital of Stomatology, Sun Yat-Sen University
Other Study IDs: GHKQ-202502-L1
Record Dates: First submitted 2025-03-07; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Maxillary Sinus Floor Elevation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Translateral: Patients undergoing translateral maxillary sinus floor elevation with simultaneous implantation in the maxillary molar region, and having successful osseointegration after 6 months.
  Interventions: Procedure: Translateral Maxillary Sinus Floor Elevation
- Hydraulic Transcrestal: Patients undergoing hydraulic transcrestal maxillary sinus floor elevation with simultaneous implantation in the maxillary molar region, and having successful osseointegration after 6 months.
  Interventions: Procedure: Hydraulic Transcrestal Maxillary Sinus Floor Elevation

INTERVENTIONS:
Procedure: Translateral Maxillary Sinus Floor Elevation — Translateral maxillary sinus floor elevation with simultaneous implantation in the maxillary molar region.
  Groups: Translateral
Procedure: Hydraulic Transcrestal Maxillary Sinus Floor Elevation — Hydraulic transcrestal maxillary sinus floor elevation with simultaneous implantation in the maxillary molar region.
  Groups: Hydraulic Transcrestal

SUMMARY:
The goal of this study is to investigate the clinical efficacy of different maxillary sinus floor elevation procedures based on maxillary sinus anatomy.

The main questions it aims to answer are:

* How does the anatomical morphology of maxillary sinus affect postoperative bone resorption?
* How to select the appropriate maxillary sinus floor elevation procedure based on maxillary sinus anatomy? Preoperative, immediate postoperative, and six-month postoperative CBCT images of patients undergoing translateral maxillary sinus floor elevation or hydraulic transcrestal maxillary sinus floor elevation will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing translateral maxillary sinus floor elevation or hydraulic transcrestal maxillary sinus floor elevation in the maxillary molar region.
* Patients undergoing maxillary sinus floor elevationwith simultaneous implantation in the maxillary molar region，and having successful osseointegration after 6 months from surgery.
* Patients having CBCT examination for preoperative, the day of surgery, and six months after surgery.
* Patients treated between January 1, 2016 and June 30, 2024.

Exclusion Criteria:

* Patients having osteointegration failure within six months after surgery.
* Refusal to participate in the study.
* Other conditions deemed unsuitable for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing maxillary sinus floor elevation with simultaneous implantation in the maxillary molar region, and having successful osseointegration after 6 months from surgery.
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Bone loss | 6 months after surgery
  The incidence of bone length, width and height gained in maxillary sinus are evaluated through CBCT imaging for preoperative, the day of surgery, and six months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Wang, Principal Investigator — Hospital of Stomatology, Sun Yat-Sen University